CLINICAL TRIAL: NCT03341052
Title: Characterization of Bile Acid Pathway in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-007060; K23DK114460 (NIH)
Record Dates: First submitted 2017-08-01; First posted 2017-11-14 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, High-Fat; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese Participants (Active Comparator): Participants will be on each diet for one week prior to collection of laboratory samples. Participants will be on their normal diet on weeks 1 and 3, on the high fat diet on week 2, and low fat diet on week 4.
  Interventions: Other: Normal Diet; Other: High Fat Diet; Other: Low Fat Diet
- Normal Weight Participants (Active Comparator): Participants will be on each diet for one week prior to collection of laboratory samples. Participants will be on their normal diet on weeks 1 and 3, on the high fat diet on week 2, and low fat diet on week 4.
  Interventions: Other: Normal Diet; Other: High Fat Diet; Other: Low Fat Diet

INTERVENTIONS:
Other: Normal Diet — The normal diet will consist of the participants' normal eating habits, and will be tracked by a food log. The participants will be on their normal diet during week 1 and week 3.
Other: High Fat Diet — The high fat diet will consist of 2700 kcal, 100g total fat (33%), 300mg cholesterol, 350g carbohydrates (52%), and 100g protein (15%). The participants will be on this diet during week 2.
Other: Low Fat Diet — The low fat diet will consist of 1200 kcal, 26g fat (20%), 78mg cholesterol, 150g carbohydrates (50%), and 100g protein (30%). The participants will be on this diet during week 4.

SUMMARY:
It is unknown whether the bile acid pathway is altered in obesity. This study is designed to compare obesity and health to determine if the bile acid pathway differs depending on health state.

DETAILED DESCRIPTION:
This is a single center study involving diet intervention, including healthy obese and healthy normal weight participants. Participants will maintain their normal diet for 1 week, eat a high fat and high calorie diet for 1 week, return to their normal diet for 1 week, and eat a low fat and low calorie diet for 1 week, to study the effect of diet on the bile acid pathway in normal weight and obesity. During their first normal diet week, the high calorie week, and the low calorie week, blood samples will be collected at defined times to measure cholesterol, glycemia, Fibroblast Growth Factor 19 (FGF-19), Bile Acid (BA), C4, and incretins (GLP-1 (glucagon-like peptide-1), peptide tyrosine tyrosine (PYY 3-36)) fasting levels and responses to the meal. Stool samples will be collected for 48 hour BA excretion.

ELIGIBILITY:
Normal Weight Inclusion Criteria:

* Women of childbearing potential will have negative pregnancy tests within 48 hours of enrollment
* BMI: 18.5-25 kg/m2

Obese Inclusion Criteria:

* Women of childbearing potential will have negative pregnancy tests within 48 hours of enrollment
* BMI: ≥ 30 kg/m2

Exclusion Criteria for both Normal Weight and Obese Participants:

* History of abdominal surgery including cholecystectomy and other than appendectomy, Caesarian section or tubal ligation.
* Positive history of chronic gastrointestinal diseases, or systemic disease that could affect gastrointestinal motility, or use of medications that may alter gastrointestinal motility, appetite or absorption, e.g., orlistat, phentermine.
* Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory (HAD), a self-administered alcoholism screening test (AUDIT-C) and the Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia). If such a dysfunction is identified by a HAD score >11 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up. The AUDIT-C is a 3-item alcohol screening questionnaire that reliably identifies participants who are hazardous alcohol drinkers or have active alcohol use disorders. In men, a score of 4 or more is above the recommended limits will be reviewed by study personnel. In women, a score of 3 or more is above the recommended limits will be reviewed by study personnel. However when the points are above recommended limits, the provider will review the patient's alcohol intake over the past few months to confirm accuracy and determine study eligibility..
* Intake of medication, whether prescribed or over the counter (except multivitamins), within 7 days of the study. Exceptions are birth control pill, estrogen replacement therapy, and thyroxin replacement therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2021-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres J Acosta Cardenas, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obese Participants | Normal Weight Participants
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Participants | Normal Weight Participants | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12) | 33 (9) | 36 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in 48h-fecal Bile Acid Excretion (μmol/L) Between Baseline and High Fat Diet
Description: Change in 48h-fecal bile acid excretion (μmol/L) between baseline and high fat diet
Time Frame: Baseline to approximately day 7 of week 2
Measure: Mean (Standard Deviation); unit: (μmol/L)/48 hour
Arm/Group | Obese Participants | Normal Weight Participants
Number analyzed (Participants) | 8 | 8
(μmol/L)/48 hour | 543 (313) | 344 (445)

2. Primary Outcome: Change in 48h-fecal Bile Acid Excretion (μmol/L) Between Baseline and Low Fat Diet
Description: Change in 48h-fecal bile acid excretion (μmol/L) between baseline and low fat diet
Time Frame: Baseline to approximately day 7 of week 4
Measure: Mean (Standard Deviation); unit: (μmol/L)/48 hour
Arm/Group | Obese Participants | Normal Weight Participants
Number analyzed (Participants) | 8 | 8
(μmol/L)/48 hour | 717.6 (666.1) | 297 (237.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 5 weeks on all participants
Groups:
- Obese: Obese
- Healthy Weight: Healthy weight
Arm/Group | Obese | Healthy Weight
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03341052/Prot_SAP_000.pdf